CLINICAL TRIAL: NCT00579397
Title: Markers of Inflammation in Hematopoietic Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Reggie E Duerst, MD, Clinical Director - Stem Cell Transplant, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: SCT 0407
Record Dates: First submitted 2007-12-21; First posted 2007-12-24 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Acute Graft Versus Host Disease
Keywords: Markers of Inflammation; acute graft versus host disease; predicting aGVHD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2.5 mL's of whole blood are obtained one time a week for the first 100 days of transplant
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: For Objective #1:
  * Healthy adult volunteers
- 2: For Objectives #2 & #3:
  * Recipients undergoing an allogeneic stem cell transplant

SUMMARY:
Objectives:

1. To show feasibility and reproducibility of performing a multiplex ligation-dependent amplification procedure (RT-MLPA)
2. To describe the profile of changes in inflammatory gene products, using RT-MLPA, in pediatric patients receiving stem cell transplant
3. To determine if changes in a specific inflammatory product, or a combination of inflammatory products, can predict grade 2-4 acute graft-versus-host disease

DETAILED DESCRIPTION:
Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) is a successful treatment option for multiple malignant diseases (i.e. leukemia) and non-malignant disorders (i.e. metabolic disorders, genetic disorders, immunodeficiencies). Unfortunately, transplantation from an HLA-related family member is only available in 30-40% of stem cell transplant recipients. The other patients requiring HSCT must then receive their stem cells from either a matched-unrelated donor (MUD) or from cord blood. One major limitation upon receiving these unrelated stem cells are acute and chronic graft-versus-host disease. Specifically looking at acute graft-versus-host disease (aGVHD), up to 30% of the recipients of stem cells from an HLA-identical related donor will develop greater or equal to grade 2 of aGVHD despite immunosuppressive prophylaxis. The percentages of patients who develop aGVHD from unrelated donors are even higher.

The current standard treatment for aGVHD is corticosteroids. Unfortunately, only 40% of matched-siblings HSCT cases and 25% of MUD SCT cases show a complete response to these steroids. Those patients who do not respond to corticosteroids can show a dismal outcome. Given the poor outcome with refractory GVHD, there has been a lot of interest in trying to predict who will get GVHD. These findings could lead to augmentation of GVHD prophylaxis.

The purpose of this study is to look at a series of identified biomarkers to predict aGVHD. Once blood is drawn from the SCT recipient, a multiplex ligation-dependent probe amplification (MLPA) will test different biomarkers in the blood to result in about 30-45 target sequences being examined simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Objective #1:
* Healthy adult volunteers, affiliated to Children's Memorial Hospital
* Male or female
* Objective #2 & #3:
* Recipient undergoing an allogeneic stem cell transplant
* Receiving related or unrelated cord blood, related or unrelated bone marrow or peripheral blood stem cells
* Any pre-transplant regimen
* Ages of 0-21 years old
* Male or female

Exclusion Criteria:

* Inability for subject/parent to understand study and therefore unable to consent
* Children under 7.0 kgs

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients undergoing a hematopoietic stem cell transplant at Children's Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2012-12-12 (Actual)

PRIMARY OUTCOMES:
To show feasibility and reproducibility of performing a multiplex ligation-dependent amplification procedure (RT-MLPA) | Until September 2008

SECONDARY OUTCOMES:
To describe the profile of changes in inflammatory gene products, using RT-MLPA, in pediatric patients receiving stem cell transplant | Until September 2008
To determine if change in a specific inflammatory product, or a combination of inflammatory products, can predict grade 2-4 acute graft-versus-host disease | Until September 2008

CONTACTS AND LOCATIONS:
Overall Officials: Reggie Duerst, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Lurie Children's Hospital, Chicago, Illinois, United States